CLINICAL TRIAL: NCT04363957
Title: Prospective, Randomized Evaluation of Patient Reported Knowledge and Satisfaction Following the Use of an Enhanced Gynecologic Brachytherapy-Specific Educational Video
Brief Title: Gynecologic Brachytherapy-Specific Educational Video
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jyoti Mayadev, MD, Associate Clinical Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 181519
Record Dates: First submitted 2020-04-03; First posted 2020-04-27 (Actual); Results first posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Cervical Cancer; Uterine Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Neoplasms

STUDY DESIGN:
Intervention Model Description: In this open-label study design, eligible participants will be randomized using a simple 1:1 schedule to either brachytherapy verbal standard consent (Arm A), or the brachytherapy specific video (Arm B), based on chronological arrival in clinic
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Consent (Other): Patients only receive the standard brachytherapy consent process
  Interventions: Other: Standard Brachytherapy Consent Process
- Standard Consent and Video Intervention (Experimental): Patients receive the standard brachytherapy consent process and the addition of an informational video about brachytherapy
  Interventions: Other: Brachytherapy video; Other: Standard Brachytherapy Consent Process

INTERVENTIONS:
Other: Brachytherapy video — Patients will watch a video that contains information about brachytherapy
  Arms: Standard Consent and Video Intervention
Other: Standard Brachytherapy Consent Process — Patients will have the standard clinical brachytherapy consent and education including discussion with their physician.

SUMMARY:
Brachytherapy is a highly technical and integral component of the definitive treatment of gynecologic cancers [1]. To enhance provider communication and patient engagement, our study investigates a video consent on impact of patient treatment-related outcomes.

The study team will use a detailed brachytherapy video in addition to the standard brachytherapy verbal consent to evaluate patient-reported satisfaction and patient anxiety for gynecologic high-dose rate brachytherapy (a radiation procedure).

DETAILED DESCRIPTION:
1:1 randomized trial using blocked randomization based on chronologic arrival in clinic, a group of patients will be randomized to the standard of care verbal consent (Arm A), or the standard of care consent plus the online brachytherapy informed video consent (Arm B). There will be three time points for the collection: After the standard consent process as the baseline, following the standard only vs standard and educational video consent process prior to the first brachytherapy procedure, and prior to the last brachytherapy procedure. The patients in the brachytherapy video consent process will be watching this online. The patient will be given a specific log in to use, and study researchers will be able to track the number of times the patient watches the video and the completion of the video view. The patient is allowed to watch the video as many times as desired

ELIGIBILITY:
Inclusion Criteria:

1. Patient has the ability to understand and the willingness to sign a written informed consent.
2. Patient must be female, all races and ethnic groups are eligible.
3. Must be > 18 years of age, or have parental approval for inclusion.
4. Must carry a diagnosis of gynecologic malignancy.
5. Is deemed to require high-dose rate gynecologic brachytherapy procedure (intracavitary, hybrid intracavitary/interstitial, or interstitial).
6. Any prior external beam radiation therapy is allowed.
7. Any performance status is allowed.
8. Women of child-bearing potential and men with partners of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for # days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

   * A woman of child-bearing potential is any female (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

     * Has not undergone a hysterectomy or bilateral oophorectomy; or
     * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)

Exclusion Criteria:

* 1. Patient has had prior high-dose rate gynecologic brachytherapy at any point in the past.

  2. . Patient is a non English speaker

  3. Patient is unable to watch the video

  4. Patient declines consent to the study

  5. Study-specific exclusion criteria.

  6. Patient has a severe or uncontrolled medical disorder that would, in the investigator's opinion, impair ability to receive study treatment (i.e., uncontrolled diabetes, chronic renal disease, chronic pulmonary disease or active, uncontrolled infection, psychiatric illness/social situations that would limit compliance with study requirements).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti Mayadev, MD, Principal Investigator — University of California, San Diego
Locations (1):
- Moores UC San Diego Cancer Center, La Jolla, California, United States

REFERENCES:
- [Derived] Kotha NV, Guram K, Morgan K, Deshler L, Brown D, Rash D, Dyer B, McHale M, Yashar C, Scanderbeg D, Einck J, Mayadev J. A randomized patient education trial investigating treatment-related distress and satisfaction with the use of an at-home gynecologic brachytherapy educational video. Int J Gynecol Cancer. 2023 Jul 3;33(7):1125-1131. doi: 10.1136/ijgc-2023-004331. PMID 37247940

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Consent | Standard Consent and Video Intervention
Started | 40 | 40
Completed | 29 | 28
Not Completed | 11 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Consent | Standard Consent and Video Intervention | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Continuous [Median (Full Range); unit: Years] | 58 [26 to 88] | 60 [32 to 89] | 59 [26 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 28 | 57
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 12
  Not Hispanic or Latino | 22 | 20 | 42
  Unknown or Not Reported | 2 | 1 | 3
Primary Cancer [Count of Participants; unit: Participants]
  Cervix | 15 | 16 | 31
  Uterine | 13 | 10 | 23
  Vagina | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Patient Reported Satisfaction
Description: Primary Analysis based on Intention-to-Treat population, defined as all individuals who were randomized to arm A or arm B. A Likert-scale study specific questionnaire (no unabbreviated scale title, Likert-scale is a general untitled tool) is used to calculate satisfaction score.
  Using the brachytherapy specific questionnaire, the study team will examine three patient reported time points for impact: baseline, after the consent process, and prior to the last brachytherapy procedure. For primary endpoint, a two-sample t-test will be used to compare differences of satisfaction scores at two time points (baseline and following consent process) between groups. The reporting scale is the following:
  Strongly disagree (1); Disagree (2); Uncertain (3); Agree (4); Strongly agree (5)
  Minimum: 1; Maximum: 5.
  Questionnaire had 12 questions. Minimum possible score is 12; Maximum possible score is 60. Higher score means higher satisfaction.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: satisfaction score at baseline
Arm/Group | Standard Consent | Standard Consent and Video Intervention
Number analyzed (Participants) | 29 | 28
satisfaction score at baseline | 54 [45 to 54] | 55 [49 to 55]

2. Secondary Outcome: Treatment Related Anxiety
Description: Satisfactory scores at three time points will be analyzed using a mixed effect model for repeated measures (MMRM) to assess satisfactory scores trajectories between two arms. The MMRM model will include terms for time, consent arm, baseline score, arm-by-time interaction, baseline score by time interaction, plus covariates that include age, stage. Time will be treated as categorical. If values of last two time points are similar, analysis of covariance model (ANCOVA) will be used to model the change in satisfactory scores. The mean of the last two time points will be calculated. That is, the after consent score (mean values) will be regressed upon baseline score and consent arms. Patient treatment-related anxiety between groups, defined as National Comprehensive Cancer Network (NCCN) distress score, are also collected at three time points and will be analyzed using the same strategy. The NCCN distress scale is from 0 (min) -10 (max) with 10 being a value that is more distress- worse.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: anxiety score at baseline
Arm/Group | Standard Consent | Standard Consent and Video Intervention
Number analyzed (Participants) | 29 | 28
anxiety score at baseline | 4 [2 to 7] | 4 [1 to 6]

ADVERSE EVENTS:
Time Frame: 1 year, 11 months
Arm/Group | Standard Consent | Standard Consent and Video Intervention
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/28
Other Adverse Events (participants affected / at risk) | 0/29 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT04363957/Prot_SAP_000.pdf